CLINICAL TRIAL: NCT00078390
Title: A Phase I/II Study of the Safety, Pharmacokinetic Interaction and Efficacy of S-3304 in Combination With Standard Therapy in Patients With Locally Advanced Non-small Cell Lung Cancer.
Brief Title: Study of S-3304 in Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0207P1421
Record Dates: First submitted 2004-02-24; First posted 2004-02-26 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer; Stage IIIA Non Small Cell Lung Cancer; Stage IIIB Non Small Cell Lung Cancer
Keywords: Lung cancer; Lung carcinoma; Non small cell lung cancer; Stage IIIA non small cell lung cancer; Stage IIIB non small cell lung cancer; NSCLC; Stage III; chemotherapy; radiation; chemoradiation; matrix metalloproteinases; neovascularization; antiangiogenesis; type IV collagenases; Unresectable locally advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neovascularization, Pathologic | interventions — S 3304

STUDY DESIGN:
Intervention Model Description: The Phase 1 part of the study will determine the tolerable dose of S-3304 in the presence of radiation and paclitaxel/carboplatin chemotherapy in a non-randomized manner.
  The Phase 2 part will compare the effect combination of S-3304 in addition to chemo-irradiation therapy to the effect of radiation and paclitaxel/carboplatin chemotherapy alone on small cell lung tumors

ARMS (2):
- S-3304 plus chemo-irradiation (Experimental): The tolerable dose of S-3304 determined in the Phase 1 part of the study will be dosed BID along with a standard of care regimen of radiation and paclitaxel/carboplatin chemotherapy
  Interventions: Drug: S-3304; Other: Chemo-irradiation
- Chemo-irradiation (Active Comparator): The standard of care regimen of radiation and paclitaxel/carboplatin chemotherapy will be administered
  Interventions: Other: Chemo-irradiation

INTERVENTIONS:
Drug: S-3304 — S-3304 will be administered at the tolerable dose BID along with chemo-irradiation
  Arms: S-3304 plus chemo-irradiation
Other: Chemo-irradiation — Standard of care chemo-irradiation

SUMMARY:
A study to measure the safety and effectiveness of S-3304 when given in combination with conventional chemo-radiation therapy in patients with locally advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
A two part study to evaluate the safety and efficacy of S-3304 in combination with standard therapy in patients with locally advanced non-small cell lung cancer. The first part of the study is a Phase I design to evaluate the maximum tolerated dose of S-3304 when given in combination with radiation and paclitaxel/carboplatin chemotherapy that is appropriate for further evaluation. The second part of the study is a randomized Phase II design to evaluate the efficacy of recommended S-3304 dose in combination with chemo-radiation.

ELIGIBILITY:
INCLUSION CRITERIA

* newly diagnosed non-small cell lung cancer of stage IIIA non-resectable or of stage IIIB without pleural effusion
* ECOG performance status 0-1
* adequate organ function
* clinically indicated and able to receive conventional chemoradiation therapy

EXCLUSION CRITERIA

* patients with prior history of cancer, other than basal cell carcinoma after appropriate treatment, or prior systemic chemotherapy treatment
* patients with other serious intercurrent illness including HIV/AIDS, or contraindicated for paclitaxel/carboplatin or thoracic irradiation treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2006-09-28 (Actual); Study Completion 2006-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Scripps Cancer Institute, La Jolla, California
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - University of Kansas Cancer Center, Kansas City, Kansas
  - VA Medical Center-East Orange (study available to veterans only), East Orange, New Jersey
  - The Cleveland Clinic, Cleveland, Ohio